CLINICAL TRIAL: NCT05878912
Title: The Effects of Obesity and Weight Loss in Heart Failure: Imaging the Obesity Paradox Using Magnetic Resonance Imaging and Spectroscopy - Heart Failure With Preserved Ejection Fraction Substudy
Brief Title: The Effect of Obesity and Weight Loss in Heart Failure With Preserved Ejection Fraction
Acronym: OWL-HFPEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 161729 (C); 15/SC/0004 (Other: Rsearch Ethics Committee); FS/CRTF/22/24293 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2023-03-15; First posted 2023-05-30 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Obesity
Keywords: Weight loss; Heart failure; Preserved ejection fraction; Obesity; Overweight; Magnetic resonance imaging
MeSH Terms: conditions — Obesity; Weight Loss; Heart Failure; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet (Experimental): Diet intervention (in addition to standard clinical care)
  Interventions: Other: Diet intervention
- Control (No Intervention): Standard clinical care only

INTERVENTIONS:
Other: Diet intervention — The diet intervention delivers a weight loss program. The main component is a total diet replacement low energy diet. The intervention includes a gradual food reintroduction phase and maintenance strategies.
  Arms: Diet

SUMMARY:
This study looks at the effects of weight loss in people who have heart failure with preserved ejection fraction (HFpEF) and are overweight or obese.

The main questions it aims to answer are whether weight loss in this group of people improves:

1. The heart's shape, how well it pumps blood and how well it uses fuels
2. The person's quality of life and how much they can exercise

Participants will attend 2 study visits, separated by 3-6 months. The intervention period takes place in between the 2 study visits.

Each study visit will involve measurements including:

* Symptom and quality of life questionnaires
* Body measurements such as height and weight
* Blood tests
* Ultrasound scans of the heart (echocardiogram)
* Magnetic Resonance Imaging (MRI) scans of the heart
* Exercise components during the scans
* 6 minute walk test

Participants are randomly allocated (in other words, by lottery) to either 'diet' or 'control' groups. The control group will continue standard care.

The diet group will be enrolled in a weight loss program supervised by the study team. Participants in the diet group will replace their usual meals with meal replacement products specifically designed to deliver a low calorie diet for weight loss. The products will consist of formula soups, shakes and porridges. This diet would last 8 weeks, followed by a guided period of food reintroduction and maintenance.

DETAILED DESCRIPTION:
An interim analysis is planned at 60 recruits to review the recruitment target.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with preserved ejection fraction (HFpEF)
* Left ventricular ejection fraction (LVEF) =/> 50%
* Body Mass Index (BMI) approximately =/> 27.5 kg/m^2

Exclusion Criteria:

* Contraindications to magnetic resonance imaging
* NYHA class IV
* Significant valvular, ischemic, infiltrative or other potentially confounding cardiac disease
* Pregnancy, planned pregnancy or lactating
* Any other conditions which may potentially compromise the safety or scientific validity of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Left atrial volume | Change from baseline at 3-6 months
  measured on cardiac magnetic resonance imaging

SECONDARY OUTCOMES:
Body weight | Change from baseline at 3-6 months
Six minute walk distance | Change from baseline at 3-6 months
N-terminal pro brain natriuretic peptide (NT pro BNP) | Change from baseline at 3-6 months
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Change from baseline at 3-6 months
  Score of 0 to 100, High scores indicate better outcome

OTHER OUTCOMES:
New York Heart Association (NYHA) class | Change from baseline at 3-6 months
  Scale from 1 to 4, Higher score indicates worse outcome
Insulin resistance | Change from baseline at 3-6 months
  Homeostatic Model Assessment for Insulin Resistance (HOMA-IR); calculated from measurements of blood glucose (millimoles per litre) and blood insulin (picomoles per litre) concentrations
Left ventricular mass | Change from baseline at 3-6 months
  calculated from volumetric analysis using cardiac magnetic resonance imaging
E/E' | Change from baseline at 3-6 months
  A measure of diastolic function on echocardiography, based on E (mitral inflow velocity) and E' (tissue doppler E' velocity)
Pulmonary artery systolic pressure | Change from baseline at 3-6 months
  On echocardiography, calculated based on tricuspid valve regurgitant velocity and estimated right atrial pressure using inferior vena cava measurement
Left atrial volume | Change from baseline at 3-6 months
  On echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Oliver J Rider, DPhil, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Clinical Magnetic Resonance Research, John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No